CLINICAL TRIAL: NCT03792594
Title: The Effect of Autologous Bone Marrow Concentration Combined With Arthroscopy for Rotator Cuff Tear
Brief Title: Autologous Bone Marrow Concentration for Rotator Cuff Tear
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Superintendent, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Other Study IDs: RD106055
Record Dates: First submitted 2019-01-02; First posted 2019-01-03 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Rotator Cuff Tear; Bone Marrow
Keywords: Bone Marrow; Mesenchymal Stromal Cells; Rotator Cuff Tear
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone marrow concentration group: The patients receive arthroscopic repair with bone marrow concentration.
  Interventions: Other: arthroscopic repair with bone marrow concentration
- Historical control group: The patients receive arthroscopic repair only
  Interventions: Other: arthroscopic repair

INTERVENTIONS:
Other: arthroscopic repair with bone marrow concentration — arthroscopic repair with bone marrow concentration
  Groups: Bone marrow concentration group
Other: arthroscopic repair — arthroscopic repair only
  Groups: Historical control group

SUMMARY:
This study aims to evaluate the effect of bone marrow concentration on healing of rotator cuff tear by comparing clinical and imaging outcomes between patients receiving arthroscopic repair with intraoperative bone marrow concentration and those receiving arthroscopic repair only.

DETAILED DESCRIPTION:
Rotator cuff tear is a common cause of pain and disability among adults. Most tears are largely caused by the normal wear and tear that goes along with aging. Although nonsurgical treatment relieves pain and improves function in the shoulder, surgical repair for a torn rotator cuff is indicated if symptoms persisted or deteriorated after 3 months nonsurgical treatments, Recently, arthroscopic repair has become the mainstream of surgical repair for rotator cuff tear. However, the healing of a repaired tendon is not always predictable. Mesenchymal stem cells (MSCs) are pluripotent cells that can differentiate into multiple mesenchymal tissues, including tenocytes, chondrocytes and osteoblasts, as well as being a source of multiple growth factors to establish an environment conducive to soft and hard tissue regeneration. As bone marrow concentration has high concentration of mesenchymal stem cells, some studies have shown that autologous bone marrow concentration can improve the healing of tendon grafts in a bone tunnel. Therefore, the goal of this study was to evaluate the effect of bone marrow concentration on healing of rotator cuff.

ELIGIBILITY:
Inclusion Criteria:

* With diagnosis of rotator cuff tear
* Age between 40 and 70 years

Exclusion Criteria:

* With prior history of shoulder surgery
* With current or prior history of trauma or infection at shoulder
* With current diagnosis of coagulopathy
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive eligible patients who underwent arthroscopic repair combined with autologous bone marrow stem cells treatment for rotator cuff tear
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-05-12 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
3-month postoperative shoulder function evaluated by Constant Shoulder Score | 3-month postoperative
  Shoulder function is evaluated using Constant Shoulder Score. The survey scores range from 0-100 with higher scores representing less dysfunction and better outcomes.

SECONDARY OUTCOMES:
6-month postoperative shoulder function evaluated by Constant Shoulder Score | 6-month postoperative
  Shoulder function is evaluated using Constant Shoulder Score. The survey scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
12-month postoperative shoulder function evaluated by Constant Shoulder Score | 12-month postoperative
  Shoulder function is evaluated using Constant Shoulder Score. The survey scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
3-month postoperative degree of healing evaluated by plain radiograph | 3-month postoperative
  Degree of healing evaluated by plain radiograph
6-month postoperative degree of healing evaluated by plain radiograph | 6-month postoperative
  Degree of healing evaluated by plain radiograph
12-month postoperative degree of healing evaluated by plain radiograph | 12-month postoperative
  Degree of healing evaluated by plain radiograph
6-month postoperative degree of healing evaluated by MRI | 6-month postoperative
  Degree of healing evaluated by MRI
12-month postoperative degree of healing evaluated by MRI | 12-month postoperative
  Degree of healing evaluated by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No